CLINICAL TRIAL: NCT06733116
Title: Standardizing Reporting Practices for Isokinetic Testing: a Delphi Study
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: INSERM UMR U1075 Comète GIP Cyceron, unicaen, Caen Normandie (Unknown)
Responsible Party: Principal Investigator, Joffrey DRIGNY, Assistant Professor, Consultant Physician, University Hospital, Caen
Other Study IDs: Delph-iso
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Developing a Consensus Framework to Standardize Isokinetic Testing Data Reporting
Keywords: isokinetic; Delphi method; strength assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group of experts in the field of isokinetic testing: A panel of experts in isokinetic testing, including physicians, physiotherapists, kinesiologists and exercise physiologists with significant expertise and recognition, will participate in a Delphi process to establish a consensus on standardizing data reporting.
  Interventions: Other: Delphi method survey

INTERVENTIONS:
Other: Delphi method survey — This intervention involves a Delphi method study, where a panel of experts in isokinetic testing will collaborate to reach a consensus on best practices for standardizing the reporting of isokinetic test data. Unlike other clinical studies, this intervention focuses on gathering expert opinions iteratively to establish a unified framework for data reporting, without direct clinical or experimental treatment. The process includes multiple rounds of feedback, refining key elements related to testing protocols, measurement parameters, and result presentation, ensuring broad expertise from various fields such as medicine, rehabilitation, and biomechanics.

SUMMARY:
Isokinetic testing plays a crucial role in research and clinical practice, particularly for evaluating muscle strength, functional performance, and imbalances between muscle groups in fields such as rehabilitation, sports medicine, and orthopedics. Despite its widespread use, there is no international consensus on how to standardize protocols or report results, leading to significant variability in methodologies, measurement parameters, and data presentation.

This Delphi method study aims to develop a consensus framework for standardizing the reporting of isokinetic testing data, ensuring consistency and comparability in research and clinical practices.

DETAILED DESCRIPTION:
Isokinetic tests are widely used in research and clinical practice to evaluate muscle strength, imbalances between muscle groups, and functional performance. These assessments are particularly important in rehabilitation, sports medicine, and orthopedics. However, the diversity in testing protocols, measured parameters, and reporting methods creates significant challenges for the comparability and interpretation of results.

Currently, there is no international consensus on how to report isokinetic test results. Scientific publications and clinical reports vary greatly in methodologies, units of measurement, and presentation of findings. Additionally, there is considerable heterogeneity in how results are presented, particularly regarding essential elements that ensure methodological reproducibility. This variability complicates the synthesis of data across studies and limits their practical application. As a result, healthcare professionals and researchers struggle to compare results, replicate studies, or effectively use the data in clinical decision-making.

The need to standardize reporting practices for isokinetic tests is therefore clear. A standardized framework would harmonize reporting, facilitate comparisons between studies, support the evaluation of therapeutic interventions, and improve the monitoring of patients or athletes over time. It would also enhance transparency and scientific rigor, which are critical for advancing knowledge and improving care.

The Delphi method, used in this study, is particularly suited to addressing this issue. It relies on an iterative process to gather the opinions of a panel of experts and establish a consensus on specific recommendations. By involving experts from various fields (physicians, physiotherapists, kinesiologists, and sport physiologists), this method ensures that the recommendations reflect a broad and balanced perspective. It also helps structure and prioritize key points, identifying essential elements for a standardized report.

The results of this study are expected to have several significant outcomes. First, they will provide a clear framework for standardizing the reporting of isokinetic tests, improving the quality and utility of the data reported. Second, this framework could be adopted internationally, fostering better collaboration between researchers and clinicians. Finally, it could serve as a foundation for developing official guidelines or recommendations, enhancing the validity and impact of isokinetic testing in clinical and scientific practices.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated knowledge or experience in isokinetic testing, such as research, clinical practice, or equipment design.
* Clinicians, researchers, educators, or professionals with relevant expertise in rehabilitation, sports medicine, biomechanics, or related fields.
* At least 5 peer-reviewed publication (first author) or equivalent contribution in the field of isokinetic testing or related domains.
* Minimum of 5 years of professional experience in a relevant field.
* Agreement to participate in all Delphi rounds and provide informed consent.
* Ability to communicate and provide responses in the language used for the study (English).

Exclusion Criteria:

* Professionals with conflicts of interest that could bias their contributions, such as direct financial ties to specific isokinetic testing equipment manufacturers.
* Inability or unwillingness to commit to the iterative Delphi process, including providing timely responses to questionnaires.
* Accidental inclusion of an expert already represented in another capacity within the study (e.g., as a member of the organizing committee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes a diverse group of experts such as physicians, physiotherapists, kinesiologists, and sport physiologists. These professionals are selected for their expertise in isokinetic testing and its application in clinical practice, rehabilitation, and sports science. The panel aims to represent a broad range of perspectives to ensure a comprehensive and standardized framework for reporting isokinetic testing data.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Consensus on Key Elements for Standardized Reporting of Isokinetic Testing | At the completion of the final Delphi round (approximately 6 months).
  The proportion of agreement among experts on the key elements to include in a standardized framework for reporting isokinetic testing data, as determined by the final round of the Delphi process. Agreement will be defined as at least 80% agreement (4 or 5 on a 5 -level Likert scale, minimum=1 maximum=5, 5 corresponding to 'strongly agree')

SECONDARY OUTCOMES:
Open Survey to Inform Delphi Rounds | At the end of the first Delphi round (approximately 2 month)
  The identification and categorization of items related to isokinetic testing, informed by an initial literature review and expert input during Round 1 of the Delphi process.
Prioritization of Reporting Items | During intermediate Delphi rounds (approximately 3-4 months).
  Ranking of reporting items by importance ("1 = optional", "2 = recommended", "3 = essential"), with 'essential' indicating that the item is mandatory, based on iterative feedback from Delphi panelists.
Years of Professional Practice | At the beginning of the Delphi process (baseline).
  Average and range of years of professional experience in fields related to isokinetic testing (e.g., sports medicine, rehabilitation, research).
Academic Contributions | At the beginning of the Delphi process (baseline).
  Number of peer-reviewed publications or other academic contributions related to isokinetic testing or related fields, self-reported by the participants.
Geographic Distribution of Expert Panel Participants | At the beginning of the Delphi process (baseline).
  Distribution of experts by geographic region (e.g., continents, countries) to evaluate the representativeness of the panel.
Expert Panel Composition - gender | At the beginning of the Delphi process (baseline).
  Analysis of gender distribution within the expert panel
Expert Panel Composition - country | At the beginning of the Delphi process (baseline).
  Analysis of the country of residence distribution within the expert panel
Expert Panel Composition - job | At the beginning of the Delphi process (baseline).
  Analysis of the type of job distribution within the expert panel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schindler IFSR, Pontes SS, Bertoni MBM, Junior GF, Junior BRN, de Jesus FLA, Neto MG. A Systematic Review of Isokinetic Muscle Strength in a Healthy Population With Special Reference to Age and Gender. Sports Health. 2023 May;15(3):328-332. doi: 10.1177/19417381221146258. Epub 2023 Jan 16. PMID 36645122
- [Background] Wilk KE, Arrigo CA, Davies GJ. Isokinetic Testing: Why it is More Important Today than Ever. Int J Sports Phys Ther. 2024 Apr 1;19(4):374-380. doi: 10.26603/001c.95038. eCollection 2024. PMID 38576833